CLINICAL TRIAL: NCT04831879
Title: Automated Mechanical Peripheral Stimulation to Treat Freezing of Gait in Patients With Parkinson's Disease and Subthalamic Nucleus Deep Brain Stimulation (STN-DBS) - a Randomized Double-blind, Sham Controlled, Cross-over Trial
Brief Title: Automated Mechanical Peripheral Stimulation to Treat Freezing of Gait in Patients With Parkinson's Disease and STN-DBS
Acronym: AMBITION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gondola Medical Technologies SA (Industry)
Collaborators: University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UKK - AMBITION
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Freezing Of Gait; FOG; Deep Brain Stimulation; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled cross-over trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A AMPS - sham (Experimental): Treatment phase 1: AMPS Treatment phase 2: sham
  Interventions: Device: GONDOLA AMPS
- Group B sham - AMPS (Experimental): Treatment phase 1: sham Treatment phase 2: AMPS
  Interventions: Device: GONDOLA AMPS

INTERVENTIONS:
Device: GONDOLA AMPS — The Gondola device is composed of two units, one per foot, each having two motors that activate rounded stimulation tips that interact with the target points. It delivers mechanical, pressure-based stimulations, sequentially in each of the four points, for the duration of 6 seconds per point. This treatment cycle is repeated 4 times, for an overall treatment duration of less than 2 minutes

SUMMARY:
The objective is to investigate whether AMPS (Automated Mechanical Peripheral Stimulation) is effective in reduction of FOG measured via the FOG-AC (Freezing Of Gait Assessment Course) in people with Parkinson Disease and STN-DBS (Subthalamic Nucleus Deep Brain Stimulation) in a randomized, double-blind, sham-controlled, cross-over trial

DETAILED DESCRIPTION:
The effects of AMPS treatment (effective vs sham) will be measured using the FOG-AC assessment. Patients will be randomized to receive either AMPS treatment and then sham or sham and then AMPS. Each treatment phase will be 4 weeks of treatment, separated by a 6-week washout period.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* ≥18 years old
* Diagnosis of Parkinson's Disease according to the United Kingdom Brain Bank Criteria
* Bilateral STN-DBS for at least 6 months
* Moderate to severe FOG i.e. FOG-AC ≥8 pts.

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Pregnancy
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* L-Dopa induced-freezing (defined by medical history),
* DBS-induced freezing (defined by medical history),
* Clinically relevant depression
* Clinically relevant cognitive impairments
* Shoe size greater than 46

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-04-27 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Freezing of gait assessment course | 4 weeks
  The primary outcome is the change in FOG severity measured by the freezing of gait assessment course (FOG-AC) and evaluated by a blinded observer using video recordings (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment).
  Min: 0 Max: 36 Higher score indicates worse symptoms.

SECONDARY OUTCOMES:
Freezing of Gait Questionnaire | 4 weeks
  FOG-Q (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment).
  Min: 0 Max: 24 Higher score indicates worse symptoms.
Timed up and go test | 4 weeks
  TUG (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment).
  Min: 16 Max: 64 Higher score indicates worse symptoms.
Movement Disorder Society - Unified Parkinson's Disease Rating Scale part I-IV | 4 weeks
  MDS-UPDRS I-IV (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment).
  Minimum score for all sections is 0, with higher scores indicating worse symptoms. Maximum value per section:
  I: 44 II: 52 III: 108 IV: 24
Parkinson's Disease Questionnaire | 4 weeks
  PDQ-39 (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment) Min: 0 Max: 100 Higher score indicates worse symptoms.
Clinical Global Impression Severity and Improvement Scores | 4 weeks
  CGI-S and CGI-I (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment).
  Min per scale: 1 Max per scale: 7 With higher score indicating worse symptoms.
Falls Efficacy Scale - International | 4 weeks
  FES-I (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment)
Fast 360° turns | 4 weeks
  Detection of freezing of gait in patients with Parkinson's disease (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment)
30-meter walk | 4 weeks
  Assessment to measure walking speed, functional mobility, gait, and vestibular function. (difference between the change after 4 weeks of effective AMPS treatment and after 4 weeks of sham-treatment)

OTHER OUTCOMES:
Parkinson Neuropsychometric Dementia Assessment | Duration of study, from screening to last follow-up visit, approximately 26 weeks
  PANDA Minimum value is 0, and the maximal raw scores of the subtests are associate learning immediate: 12, ﬂuency: no maximum, working memory: 6, spatial imagery: 3, associate learning delayed: 4. Higher score indicate lesser symptoms.
Beck's Depression Inventory | Duration of study, from screening to last follow-up visit, approximately 26 weeks
  BDI Min per scale: 0 Max per scale: 63 With higher score indicating worse symptoms.
Levodopa equivalent daily dose | Throughout the duration of study, approximately 26 weeks
  LEDD
Deep Brain Stimulation - Total Electrical Energy Delivered | Throughout the duration of study, approximately 26 weeks
  DBS TEED

CONTACTS AND LOCATIONS:
Overall Officials: Michael Barbe, MD, Principal Investigator — Department of Neurology, University Hospital Cologne
Locations (1):
- Uniklinik Köln, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Stocchi F, Sale P, Kleiner AF, Casali M, Cimolin V, de Pandis F, Albertini G, Galli M. Long-term effects of automated mechanical peripheral stimulation on gait patterns of patients with Parkinson's disease. Int J Rehabil Res. 2015 Sep;38(3):238-45. doi: 10.1097/MRR.0000000000000120. PMID 26164797
- [Background] Quattrocchi CC, de Pandis MF, Piervincenzi C, Galli M, Melgari JM, Salomone G, Sale P, Mallio CA, Carducci F, Stocchi F. Acute Modulation of Brain Connectivity in Parkinson Disease after Automatic Mechanical Peripheral Stimulation: A Pilot Study. PLoS One. 2015 Oct 15;10(10):e0137977. doi: 10.1371/journal.pone.0137977. eCollection 2015. PMID 26469868
- [Background] Prusch JS, Kleiner AFR, Salazar AP, Pinto C, Marchese RR, Galli M, Pagnussat AS. Automated mechanical peripheral stimulation and postural control in subjects with Parkinson's disease and freezing of gait: a randomized controlled trial. Funct Neurol. 2018 Oct/Dec;33(4):206-212. PMID 30663967
- [Background] Pinto C, Pagnussat AS, Rozin Kleiner AF, Marchese RR, Salazar AP, Rieder CRM, Galli M. Automated Mechanical Peripheral Stimulation Improves Gait Parameters in Subjects With Parkinson Disease and Freezing of Gait: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2018 Jun;97(6):383-389. doi: 10.1097/PHM.0000000000000890. PMID 29309313
- [Background] Pagnussat AS, Salazar AP, Pinto C, Redivo Marchese R, Rieder CRM, Alves Filho JO, Franco AR, Kleiner AFR. Plantar stimulation alters brain connectivity in idiopathic Parkinson's disease. Acta Neurol Scand. 2020 Sep;142(3):229-238. doi: 10.1111/ane.13253. Epub 2020 May 5. PMID 32299120
- [Background] Pagnussat AS, Kleiner AFR, Rieder CRM, Frantz A, Ehlers J, Pinto C, Dorneles G, Netto CA, Peres A, Galli M. Plantar stimulation in parkinsonians: From biomarkers to mobility - randomized-controlled trial. Restor Neurol Neurosci. 2018;36(2):195-205. doi: 10.3233/RNN-170744. PMID 29526852
- [Background] Kleiner AFR, Souza Pagnussat A, Pinto C, Redivo Marchese R, Salazar AP, Galli M. Automated Mechanical Peripheral Stimulation Effects on Gait Variability in Individuals With Parkinson Disease and Freezing of Gait: A Double-Blind, Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Dec;99(12):2420-2429. doi: 10.1016/j.apmr.2018.05.009. Epub 2018 Jun 11. PMID 29902470
- [Background] Kleiner A, Galli M, Gaglione M, Hildebrand D, Sale P, Albertini G, Stocchi F, De Pandis MF. The Parkinsonian Gait Spatiotemporal Parameters Quantified by a Single Inertial Sensor before and after Automated Mechanical Peripheral Stimulation Treatment. Parkinsons Dis. 2015;2015:390512. doi: 10.1155/2015/390512. Epub 2015 Oct 1. PMID 26495152
- [Background] Galli M, Vicidomini C, Rozin Kleiner AF, Vacca L, Cimolin V, Condoluci C, Stocchi F, De Pandis MF. Peripheral neurostimulation breaks the shuffling steps patterns in Parkinsonian gait: a double blind randomized longitudinal study with automated mechanical peripheral stimulation. Eur J Phys Rehabil Med. 2018 Dec;54(6):860-865. doi: 10.23736/S1973-9087.18.05037-2. Epub 2018 Feb 19. PMID 29457707
- [Background] Barbic F, Galli M, Dalla Vecchia L, Canesi M, Cimolin V, Porta A, Bari V, Cerri G, Dipaola F, Bassani T, Cozzolino D, Pezzoli G, Furlan R. Effects of mechanical stimulation of the feet on gait and cardiovascular autonomic control in Parkinson's disease. J Appl Physiol (1985). 2014 Mar 1;116(5):495-503. doi: 10.1152/japplphysiol.01160.2013. Epub 2014 Jan 16. PMID 24436294
- [Background] Zamuner AR, Shiffer D, Barbic F, Minonzio M, Andrade CP, Corato M, Lalli S, Dipaola F, Cairo B, Albanese A, Porta A, Furlan R. Mechanical somatosensory stimulation decreases blood pressure in patients with Parkinson's disease. J Hypertens. 2019 Aug;37(8):1714-1721. doi: 10.1097/HJH.0000000000002084. PMID 31107357
- See also: Sponsor website — https://www.gondola-medical.com/